CLINICAL TRIAL: NCT01003457
Title: Ultrasonographic Bladder Wall Thickness and Different Forms of Detrusor Overactivity
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Other Study IDs: uninsubria1
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Detrusor Overactivity
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- detrusor overactivity
  Interventions: Other: ultrasonography

INTERVENTIONS:
Other: ultrasonography — transvaginal ultrasonography of bladder wall thickness

SUMMARY:
In the last decade, several authors proposed ultrasound measurement of Bladder wall thickness (BWT) for the screening of the voiding dysfunction and of the detrusor overactivity (DO). The aims of the investigator prospective study were:

* to compare the ultrasonographic measurement of BWT in women with DO vs women with other urodynamic diagnosis in a very large population.
* to verify whether the BWT in women with DO can be different in the clinically or urodinamically different forms of DO.

ELIGIBILITY:
Inclusion Criteria:

* All women referred to our Urogynecology Unit from January 2005 to December 2008 for symptoms of OAB, stress urinary incontinence or mixed incontinence and sottoposte a prove urodinamiche complete were included in this prospective study

Exclusion Criteria:

* The investigators excluded women with documented recurrent urinary tract infections
* Previous antimuscarinic treatment
* Previous pelvic surgery
* Neurological disease
* Vaginal prolapse > I stage
* Symptoms or clinical and/or urodynamic signs of voiding dysfunction
* Patients included in other ongoing clinical trials during the same study period.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all women with urinary dysfunction
Sampling Method: Non-Probability Sample
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Insubria, Varese, varese, Italy

REFERENCES:
- [Derived] Serati M, Salvatore S, Cattoni E, Soligo M, Cromi A, Ghezzi F. Ultrasound measurement of bladder wall thickness in different forms of detrusor overactivity. Int Urogynecol J. 2010 Nov;21(11):1405-11. doi: 10.1007/s00192-010-1194-1. Epub 2010 Jun 10. PMID 20535449